CLINICAL TRIAL: NCT05313932
Title: The Effects of Partial Sleep Restriction on Physiological and Perceptual Responses During Submaximal and Maximal Exercise in Trained Runners
Brief Title: The Effects of Sleep Deprivation on Physiological and Perceptual Responses During Exercise
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St Mary's University College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: StMarysUC4
Record Dates: First submitted 2022-03-29; First posted 2022-04-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Sleep Deprivation
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep deprivation (Experimental): Two hours of sleep deprivation (Six hours of sleep)
  Interventions: Other: Sleep deprivation
- No intervention (No Intervention): No sleep deprivation (Eight hours of sleep)

INTERVENTIONS:
Other: Sleep deprivation — Participants wake after six hours so that they are deprived of 2 hours of sleep
  Arms: Sleep deprivation

SUMMARY:
Sleep deprivation has been found to impact exercise performance. The effects of both partial (several hours) and full (24+ hours) sleep deprivation on exercise performance has shown effects on rating of perceived exertion, rate of oxygen consumption, respiratory exchange ratio, and heart rate. A common practice with athletes is to perform regular physiological testing (submaximal and maximal) in order to assess their fitness and to determine training intensities. However, the effects of sleep deprivation on those same physiological test results has not been investigated Therefore, the purpose of this study is to investigate the effects of partial sleep deprivation on physiological test results.

ELIGIBILITY:
Inclusion Criteria:

* Injury-free, trained, male runners

Exclusion Criteria:

* Female, untrained, injured

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-04-20 (Estimated); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-09-26 (Estimated)

PRIMARY OUTCOMES:
Oxygen uptake | From baseline to completion, up to 31 days
  Change from baseline in oxygen uptake measured breath-by-breath using an online gas analyzer during submaximal and maximal incremental exercise
Respiratory exchange ratio | From baseline to completion, up to 31 days
  Change from baseline in respiratory exchange ratio measured breath-by-breath using an online gas analyzer during submaximal and maximal incremental exercise
Breathing frequency | From baseline to completion, up to 31 days
  Change from baseline in breathing frequency measured breath-by-breath using an online gas analyzer during submaximal and maximal incremental exercise
Minute ventilation | From baseline to completion, up to 31 days
  Change from baseline in minute ventilation measured breath-by-breath using an online gas analyzer during submaximal and maximal incremental exercise
Blood lactate concentration | From baseline to completion, up to 31 days
  Change from baseline in blood lactate concentration measured using capillary puncture during submaximal and maximal incremental exercise
Rating of perceived exertion | From baseline to completion, up to 31 days
  Change from baseline in ratings of perceived exertion measured using a 15-point (6-20) scale during submaximal and maximal incremental exercise
Heart rate | From baseline to completion, up to 31 days
  Change from baseline in heart rate measured using a heart rate monitor during submaximal and maximal incremental exercise

IPD SHARING:
Plan to Share IPD: No